CLINICAL TRIAL: NCT00733395
Title: Comparison of Two Juice Drinks in Preventing the Symptoms of Muscle Pain Among Runners
Brief Title: Hood to Coast Injury Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerry Kuehl, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: e4652
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: Muscle pain
MeSH Terms: conditions — Pain; Myalgia | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tart cherry juice
  Interventions: Dietary Supplement: Tart Cherry Juice
- 2 (Placebo Comparator): Fruit juice
  Interventions: Dietary Supplement: Fruit juice

INTERVENTIONS:
Dietary Supplement: Tart Cherry Juice — Participants will ingest 10.5 fl oz of cherry juice twice a day for 7 days prior to the race, and the day of the race (8 days total).
  Other Names: Cherrish
  Arms: 1
Dietary Supplement: Fruit juice — Participants will ingest 10.5 fl oz of fruit juice twice a day for 7 days prior to the race, and the day of the race (8 days total), which will serve as a 'placebo' juice.
  Arms: 2

SUMMARY:
The purpose of this study is to examine how certain kinds of fruit juice that contain natural antioxidants and natural anti-inflammatory properties may reduce exercise-induced muscle pain and injury. Participants will be recruited from registered participants in the Hood To Coast Relay. The Hood To Coast Relay Race Officials will post the study on their website to find interested teams. Interested participants will then be contacted by the study staff by phone regarding the study's inclusion and exclusion criteria and to schedule the initial health screening visit. The participants will undergo an initial health screening and survey about muscle soreness, and then drink the investigational juice twice daily for 8 days. On the 7th day of drink administration, the participants will report to the starting location of the Hood To Coast Relay to meet with the investigators for 30 minutes to survey muscle pain and juice tolerability. The participants will then participate in the Hood To Coast Relay, drinking 2 more bottles of juice over the duration of the relay. At the conclusion of the relay, the participants will meet with study investigators to take the same short survey about muscle pain and juice tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness not to take any anti-inflammatory or pain relieving drugs during the course of the study, and not to seek any other treatment for any symptoms of muscle damage until completion of the study after the race.

Exclusion Criteria:

* The investigators will exclude individuals who have or are using antiepileptic drugs for pain, acupuncture, or transcutaneous electrical nerve stimulation within 3 weeks before enrollment
* Recent use (within 5 half-lives) of topical medications/anesthetics, muscle relaxants, tender point anesthetic injections within 2 months, systemic steroids within 3 months or any investigational drug/device in the prior 30 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The administration of tart cherry juice will reduce the symptoms of exercise-induced muscle damage as measured by patients assessment of pain on a standard VAS. | Post Race

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, Principal Investigator — Oregon Health and Science University